CLINICAL TRIAL: NCT03735914
Title: Cryoneurolysis of Arnold's Nerve and Follow-up by Tractography: Feasibility Study
Acronym: CRYOARNOLD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion period finished
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC16.242
Record Dates: First submitted 2018-10-25; First posted 2018-11-08 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Neuralgia Arnold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neuralgic patients (Experimental): MRI experimentation
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Neuralgic patients for which a cryoneurolysis has been indicated, will passed an MRI befor and after the cryoneurolysis to check the presence of the nerve.

SUMMARY:
According to the World Health Organization (WHO), headaches are one of the most common nervous system disorders. The therapeutic strategy is well established for certain subcategories of headache. On the other hand, when headaches become refractory, some nerves may become the target of targeted therapies. This is the case of the Arnold nerve, also called the great occipital nerve, which is involved in certain pathologies, both physiopathologically and therapeutically. The Arnold nerve infiltration has a relatively short duration of effectiveness (about 1 month on average), some teams have reported the interest of achieving a destruction of the Arnold nerve by radio frequency, with extended durations of efficiencies to several months. The use of cryoneurolysis has been known for a long time and its effectiveness in the management of cranio-facial pain is already reported. It is thus possible to obtain, at the end of the cryoanalgesia needle, very low temperatures around -40 ° C, which leads to the formation of an ice cube and, where appropriate, the freezing of the structures (nerves among others) to the needle contacts. This induces the formation of microcrystals leading to irreversible lesions of vasa-nervorums resulting in an endoneural edema. In the long run, it appears a Wallerian degeneration without destruction of this endoneurum. This is associated with the lack of destruction of the structure of the Schwann cell. Nerve regeneration is possible.

The diffusion MRI study allows tractographic reconstruction of the nerves. This is the only imaging technique that focuses on the fibrillar structure of the nerves, thus enabling the detection of nerves throughout its path. It is a morphological imaging technique nevertheless it also allows a quantitative analysis of the nerve through certain parameters.

The Investigators hypothesize that the cryoneurolysis of the Arnold nerve will result in the disappearance of visualization of the nerve by MRI tractography. The effect of cryoneurolysis on Arnold nerves, as on other peripheral nerves through diffusion MRI has never been described. The follow-up of MRI patients who had undergone cryoneurolysis would make it possible to study the behavior of these nerves after cryoneurolysis, and to correlate the aspect in tractography with the clinical data. Painful recurrence can then be correlated with visualization of the nerves by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient with cephalalgic syndrome> 3 months,
* Patient with an indication of first cryoneurolysis
* Unilateral character of cephalalgic syndrome
* Failure of oral treatment of stage II
* Positive response (> 50% efficacy on pain EVA) to infiltration of Arnold's nerve
* Subject having signed his written participation consent

Exclusion Criteria:

* Coagulation disorder
* Infection in progress
* Patient under anticoagulant
* Contraindication to performing an MRI:

  1. Any subject with a vascular stent implanted less than 6 weeks before the examination.
  2. Any subject with implanted biomedical material deemed "unsafe" or "unsafe" in the list: http://www.mrisafety.com/TheList_search.asp.
  3. Any acquisition procedure that does not meet the conditions required for "conditional" use in a subject carrying implanted biomedical material deemed "conditional" in the list: http://www.mrisafety.com/TheList_search.asp.
  4. Any subject carrying an intra-ocular or intra-cranial ferromagnetic foreign body close to the nerve structures.
  5. Any subject carrying a biomedical material such as a cardiac, neuronal or sensory stimulator (cochlear implant) or a ventricular bypass valve without medical and paramedical supervision trained to perform MRI in these subjects.
  6. Non-cooperating subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Morphological effect of Arnold's nerve cryoneurolysis | one month
  Visualization of Arnold's nerve after tracer cryoneurolysis by MRI

SECONDARY OUTCOMES:
analgesic efficacy of the cryoneurolysis of Arnold's nerve :Measure of pain with a numeric pain scale between 0 (no pain) to 10 (intolerable) | day 7, one month, 3 months, 6 months, 12 months
  Measure of pain with a numeric pain scale between 0 (no pain) to 10 (intolerable)
Functional Impact of Pain-Related Disability After Cryoneurolysis by the Pain Disability Index Scale | day 7, one month, 3 months, 6 months, 12 months
  Score in Pain Disability Index Scale. This scale measure the interference of pain on daily activities. There are 7 items with score range from 0 (no disability) to 10 (maximum disability)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France